CLINICAL TRIAL: NCT00677716
Title: Open-label, Dose Confirmation Study of Interstitial 131I-chTNT-1/B MAb (Cotara®) for the Treatment of Glioblastoma Multiforme (GBM) at First Relapse
Brief Title: Dose Confirmation Study of Cotara for the Treatment of Glioblastoma Multiforme at First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0503
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma multiforme; GBM; brain cancer; Cotara; radioactive isotope; monoclonal antibody; Glioblastoma multiforme at first relapse
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — 131I-chimeric TNT-1-B monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131I-chTNT-1/B MAb (Cotara) (Experimental)
  Interventions: Drug: 131I-chTNT-1/B MAb (Cotara)

INTERVENTIONS:
Drug: 131I-chTNT-1/B MAb (Cotara) — Given as a single interstitial infusion over approximately 25 hours at a dose of 2.5 mCi/cc.
  Other Names: Cotara®

SUMMARY:
Cotara® is an experimental new treatment that links a radioactive isotope (iodine 131) to a targeted monoclonal antibody. This monoclonal antibody is designed to bind tumor cells and deliver radiation directly to the center of the tumor mass while minimizing effects on normal tissues. Cotara® thus literally destroys the tumor "from the inside out". This may be an effective treatment for glioblastoma multiforme, a malignant type of brain cancer.

DETAILED DESCRIPTION:
To confirm the safety and tolerability of the Maximum Tolerated Dose (MTD) of 131I-chTNT-1/B MAb given as a single interstitial infusion in patients with glioblastoma multiforme at first relapse.

To estimate overall survival, progression free survival and proportion of patients alive at six months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM
* Clinical Target Volume between 5 and 60 cc (inclusive)
* 18 to 75 years old (inclusive)
* Karnofsky Performance Status ≥ 70 percent
* If on steroids dose (± 4mg/day) must be stable for at least two weeks prior to screening/baseline visit. If not on steroids for two weeks prior to screening/baseline visit are allowed
* Adequate hematology
* Adequate renal function
* Adequate liver function

Exclusion Criteria:

* Infratentorial tumor(s), tumor(s) that communicate with the ventricles or intraventricular disease
* Bilateral non-contiguous gadolinium enhancing tumor
* Diffuse disease (i.e., any satellite lesions less than 1.5 cm from anticipated location of any catheter tip or less than two satellite lesions)
* Known or suspected allergy to study medication or iodine
* Surgical procedure within four weeks of baseline
* More than one prior chemotherapy regime or chemotherapy within four weeks (nitrosourea-based within six weeks) of baseline
* Radiation therapy within four weeks of baseline
* Investigational agent within last 30 days
* Previous treatment with any chimeric monoclonal antibody
* HIV positive
* Evidence of active hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-07; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To confirm the safety and tolerability of the maximum tolerated dose

SECONDARY OUTCOMES:
To estimate overall survival, progression free survival and proportion of patients alive at six months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak K Gupta, MBBS,MS,MCh, Principal Investigator — All India Institute of Medical Sciences
Locations (7):
- United States (3):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Pennsylvania, Department of Neurosurgery, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- India (4):
  - Amrita Institute of Medical Sciences and Research Center,, Kochi, Kerala
  - Manipal Institute for Neurological Disorders,, Bangalore
  - Department of Neurosurgery Jaslok Hospital and Research Centre, Mumbai
  - All India Instutite of Medical Sciences, New Delhi